CLINICAL TRIAL: NCT07036822
Title: Effects of Skeletal Anchored Maxillary Expander for Constricted Maxilla With Different Patient's Age (Cone Beam Computed Tomography Study)
Brief Title: Effects of Skeletal Anchored Maxillary Expander for Constricted Maxilla
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samar Hassan Mahmoud Mohamed (Other)
Responsible Party: Sponsor-Investigator, Samar Hassan Mahmoud Mohamed, Master's student, Faculty of Dental Medicine ,AL-Azhar University ,Assuit branch, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Skeletal maxillary expansion
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Maxillary Expansion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adolescent group (Experimental)
  Interventions: Device: Skeletal Anchored Maxillary Expander (MARPE)
- Adult group (Experimental)
  Interventions: Device: Skeletal Anchored Maxillary Expander (MARPE)

INTERVENTIONS:
Device: Skeletal Anchored Maxillary Expander (MARPE) — Mini implant assisted rapid maxillary expander (MARPE) used for skeletal maxillary expansion in adolescent and adult patients

SUMMARY:
The aim of study will be Evaluation of Effects of skeletal anchored maxillary expander for constricted maxilla with different patient's age

DETAILED DESCRIPTION:
Various factors contribute to transverse deficiencies in the dental arch, which can present in several ways, including posterior crossbite, a collapsed maxillary arch, discrepancies in transverse dental arch, and cleft palate. Several devices and orthopedic approaches have been developed to address transverse maxillary constriction, which can be either surgical or non-surgical, and these devices may be either fixed or removable. Various types of anchorage can be utilized, such as tooth-borne anchorage with a hyrax or tooth-tissue-borne and bone-borne methods like mini-implant-assisted rapid palatal expander (MARPE). Rapid maxillary expansion (RME) is a frequently employed and dependable technique to rectify transverse maxillary deficiencies in prepubertal and adolescent individuals. RPE successfully treats both unilateral and bilateral buccal crossbites by expanding the maxilla by separating the midpalate suture. It works especially well for developing individuals with mixed dentition, but in older teenagers, it might cause side effects such buccal tilting of teeth and periodontal issues In post pubertal individuals (including young adults and adults), the use of rapid maxillary expansion (RME) techniques remains debated, as the median palatal suture is frequently matured and challenging to open clinically. As a result, these methods might lead to negative side effects, such as dentoalveolar compensation and adverse dental and periodontal outcomes in the affected teeth instead of genuine skeletal expansion.

Mini implant-assisted rapid maxillary expansion aims to achieve skeletal expansion of the palatal arch while minimizing the unwanted dental complications The Mini screw-assisted rapid palatal expansion, designed by Lee et al., functions as a tooth-bone-borne RPE-Hyrax device that is anchored in the palate with four Mini screws connected through helical loops that were soldered to the base of the expansion screw. These tiny screws were essential in allowing the midpalatal sutures to separate by applying the expansion force straight to the palate. MARPE is employed in both adolescents and adults as an alternative to surgically assisted rapid palatal expansion (SARPE). CBCT images showed an increase in skeletal dimensions in adult and adolescent patients treated with MARPE and a reduction in dental side effects. In recent years, Mini screw-assisted rapid palatal expansion (MARPE) has emerged as a highly effective method for achieving skeletal expansion of the maxilla in adolescents and adults, especially in cases where traditional rapid palatal expansion (RPE) may be limited due to increased suture interdigitation with age. MARPE enables orthopedic expansion without the need for surgical assistance in many cases The accuracy, adaptability, and efficiency of MARPE devices have significantly increased with the incorporation of 3D printing technology. Cone-beam computed tomography (CBCT) data and digital intraoral scans are used to construct 3D-printed MARPE appliances, enabling patient-specific designs that maximize comfort, fit, and biomechanical efficacy. Mini screw placement accuracy, better appliance adaptation to palate anatomy, and less chairside time are all made possible by the digital workflow.

The present trend in orthodontics toward individualized and technologically advanced treatment options is best illustrated by the combination of MARPE and 3D printing. By providing a more pleasant and effective treatment mode, this innovation not only improves clinical outcomes but also the patient experiences

.

ELIGIBILITY:
Inclusion Criteria:

* Skeletal maxillary transverse deficiency.
* Unilateral or bilateral posterior crossbite. .Patient maintains good oral hygiene and overall health.
* Patient with no previous orthodontic treatment.
* No systemic disease that may affect bone quality or interfere with orthodontic treatment.
* Adolescent and adult patien

Exclusion Criteria:

* Craniofacial congenital disorders, including cleft lip and palate.
* History of periodontal disease

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Skeletal and dental changes after skeletal anchored maxillary expander for constricted maxilla in adolescent and adult patients constricted maxilla in adolescent and adult patients | from baseline (T0) to post expansion (T1)approximately 3 months
  changes in maxillary skeletal and dental arch width assessed by CBCT imaging before and after MARPE treatment.. evaluation includes skeletal expansion and transverse dental arch changes

CONTACTS AND LOCATIONS:
Overall Officials: Saleh Anwar Saleh, Professor of orthodontics, Study Director — ALAzhar university ,faculty of dentistry; Esmail Kamal Hewy, lecturer of orthodontics, Principal Investigator — ALAzhar university ,faculty of dentistry

IPD SHARING:
Plan to Share IPD: No